CLINICAL TRIAL: NCT03470012
Title: Adhesive Tape Trauma Evaluation of a New Gentle Tape in Healthy Infant Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-014050
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Skin (FLACC Scores of Test Subjects) After Tape Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Investigational tape
  Interventions: Device: Multi-Purpose Gentle Tape

INTERVENTIONS:
Device: Multi-Purpose Gentle Tape — The Multi-Purpose Gentle Tape is a general purpose medical adhesive tape for medical applications used primarily to secure dressings, lightweight tubing, and devices to skin.

SUMMARY:
The objective of this study is to determine the relative gentleness of a new medical tape.

DETAILED DESCRIPTION:
The objective of this study is to determine the relative gentleness of a new medical tape. A three-prong multidimensional evaluation consisting of expert grader, subject discomfort assessment, and laboratory assessments was used. One pre-study visit took place up to 7 days prior to the start of the study. The study was conducted over two days with one tape sample applied and removed. Assessments were taken on the final day. This was to mimic a normal tape application in health care practice.

ELIGIBILITY:
Inclusion Criteria: Subjects will be infants or children of either gender who meet the following criteria:

1. Who are healthy and who have intact skin at the test site with a baseline score of 0 for erythema
2. Who are between the ages of 6 months - 4 years of age (48 months)
3. Who have a Fitzpatrick Skin Type of I, II or III
4. Whose parent or legal representative agrees to not use any products (i.e. topical medications, creams, powders or ointments) on the test sites for 24 hours prior to the study start date
5. Whose parent or legal representative agrees to sponge bathe their child during the study but agrees to not bathe their child 1 hour before each visit.
6. Whose parent or legal representative agrees to not soak the tape during a sponge bath. If the site gets wet, parent or legal representative agrees to pat their child's back dry (no rubbing).
7. Whose parent or legal representative is willing to sign the Informed Consent Form (with photo release) and HIPAA Authorization.

Exclusion Criteria:

1. Who are known to be developmentally delayed
2. Who have any known allergy or sensitivity to tapes
3. Who have sunburn, skin infection or scars, moles, or other blemishes on the back that would obscure grading of the test site
4. Who have had any exposure to other topical medications, creams, powders, or ointments on the test sites 24 hours prior to the start of the study
5. Who have had a strep infection within the 2 weeks prior to the start of the study
6. Who have a history of uncontrolled diabetes, psoriasis, any active dermatitis, or recent history of dermatitis or skin reactions
7. Has participated in any study in the last 2 weeks, or are currently participating in another study, or are scheduled to participate in another study during this study period.
8. Has any other skin disorders that, in the opinion of the investigator, will interfere with the study results or will increase undue risk for the child.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Grove, PhD, Principal Investigator — Study Investigator
Locations (1):
- cyberDERM, inc., Broomall, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred between 1/16/2018 and 1/23/2018.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 27.17 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: The Face, Legs, Activity, Cry, Consolability (FLACC) Score.
Description: The Face, Legs, Activity, Cry, Consolability (FLACC) scale is a measurement used to assess pain for children Participants between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. Lower values represent lessening pain on the scale. At the 24 hour visit , a baseline FLACC score was recorded with the tape still in place. The tape was then removed and a FLACC score was recorded after removal. The reported value is the difference between FLACC after removal and FLACC at baseline.
Time Frame: 24 Hours after initial tape application and after tape removal. Change in FLACC score between the time of tape removal and baseline.
Population: Measure change in FLACC score for 24 Participants at the time of tape removal and baseline.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 24
units on a scale | 0.29 [0 to 10]

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
Relatively small sample size and no comparator product. Hard to evaluate responses of infants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03470012/Prot_SAP_000.pdf